CLINICAL TRIAL: NCT00318630
Title: A Randomised Double-blind Two-period Crossover Study to Investigate the Effect of Treatment With Repeat Doses of a PPAR Gamma Agonist on the Allergen-induced Late Asthmatic Response in Subjects With Mild Asthma Compared With Repeat Doses of Placebo
Brief Title: The Effect Of AVANDIA On The Late Asthmatic Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 104385
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Asthma AVANDIA Inflammation
MeSH Terms: conditions — Asthma | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving treatment 1 (Experimental): Eligible subjects will receive rosiglitazone immediate release tablet with a dose of 4 milligrams twice daily administered orally for 28 days followed by placebo oral tablet.
  Interventions: Drug: Rosiglitazone; Drug: Placebo
- Subjects receiving treatment 2 (Experimental): Eligible subjects will receive placebo oral tablet followed by rosiglitazone immediate release tablet with a dose of 4 milligrams twice daily for 28 days.
  Interventions: Drug: Rosiglitazone; Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone will be given as immediate release tablet of 4 milligrams administered orally for 28 days.
Drug: Placebo — Subjects will also receive placebo oral tablet.

SUMMARY:
This study is to investigate the effects of AVANDIA on the asthmatic response.

ELIGIBILITY:
Inclusion criteria:

* Mild asthmatic treated with short-acting beta agonists only, non-smoker.

Exclusion criteria:

* Inability to abstain from medications other than short-acting beta agonists and paracetamol.
* Recent administration of steroids.
* Recent respiratory infection or exacerbation of asthma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2005-07-22 (Actual); Primary Completion 2006-06-30 (Actual); Study Completion 2006-06-30 (Actual)

PRIMARY OUTCOMES:
The effect of repeat oral doses of AVANDIA for 28 days on the late asthmatic response to inhaled allergen. Measured as lung function 4-10 hours after allergen challenge after 28 days dosing. | Up to 43 days

SECONDARY OUTCOMES:
The early asthmatic response to allergen, bronchial challenge, nitric oxide, markers of inflammation and safety/tolerability. | Up to 43 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- [Derived] Richards DB, Bareille P, Lindo EL, Quinn D, Farrow SN. Treatment with a peroxisomal proliferator activated receptor gamma agonist has a modest effect in the allergen challenge model in asthma: a randomised controlled trial. Respir Med. 2010 May;104(5):668-74. doi: 10.1016/j.rmed.2009.11.006. Epub 2009 Nov 26. PMID 19944580
- See also: Results for study 104385 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/104385?search=study&search_terms=104385#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104385 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register